CLINICAL TRIAL: NCT04010591
Title: The Measurement of Bladder Impedance and Heart Rate During Urodynamic Study - Prospective Study
Brief Title: The Measurement of Bladder Impedance and Heart Rate During Urodynamic Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0500
Record Dates: First submitted 2019-04-30; First posted 2019-07-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Voiding Dysfunction
Keywords: Pediatric patients; Voiding Dysfunction; urodynamic study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UDS group: All enrolled patients with urodynamic study
  Interventions: Device: impedance measurement during urodynamic study

INTERVENTIONS:
Device: impedance measurement during urodynamic study — Impedance information is measured through the belt in the abdomen of the subject. The urodynamic test is performed from the state in which the urine of the bladder is completely emptied to the state of the bladder until the state becomes full, so the impedance measurement is measured from the state where the urine of the bladder is completely emptied to the state of the bladder until the state becomes full.

SUMMARY:
Purpose To measure the impedance of the bladder during the urodynamic study to see if changes in the impedance value occur as the bladder volume changes in pediatric patients aged 5-12 years along with its leg time.

In addition, during the urodynamics test, the heart rate is measured at the same time to confirm the pulse change due to the filling of the bladder.

-Background of the study (Method of identifying urinary bladder using impedance) In order to overcome the limitation of the method of checking the urinary volume in the bladder using ultrasound, the measurement of the impedance in the bladder is proposed as an alternative. Impedance measurement is non-invasive, very low cost, easy to measure and has a great advantage that it can be continuously measured in everyday life. In fact, early studies suggest that impedance measurement in the bladder is helpful in identifying urinary bladder capacity.

On the other hand, there are two disadvantages to the urinary bladder identification method using impedance. One is the relative aspect that the impedance value changes according to the patient, and the other is the time lag time from the measurement point to the point when the impedance change appears.

* In order to overcome this problem of impedance-based urinary bladder identification method, we measured impedance change according to real-time change of urinary volume in bladder during urodynamic study.
* Background of the Invention (Pulse changes due to changes in urinary volume in bladder) It is known that when the urine enters the urinary bladder, the autonomic nervous system detects and regulates the heart rhythm, and the change of heart rate has not been reported in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children aged 5-12 years
* 2. Children in whom urodynamic evaluation is required due to voiding dysfunction
* 3. Children who agreed to participate in clinical trials

Exclusion Criteria:

* 1. If there is a previous history of bladder surgery
* 2. If there is a scar on the upper part of the pubic bone

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Bladder Impedance | Measure the baseline before starting the inspection.
  This study was a prospective observational study of 33 patients. Impedance before the bladder filling will be measured.
Bladder Impedance | Measure up to 5 minutes after of the inspection.
  This study was a prospective observational study of 33 patients. Impedance after the bladder filling will be measured.
Bladder pulses | Measure the baseline before starting the inspection.
  This study was a prospective observational study of 33 patients. Pulses before the bladder filling will be measured.
Bladder pulses | Measure up to 5 minutes after of the inspection.
  This study was a prospective observational study of 33 patients. Pulses after the bladder filling will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No